CLINICAL TRIAL: NCT00572624
Title: Effect of Weight Loss on Myocardial Oxygen Consumption and Left Ventricular Relaxation in Obese Adults
Brief Title: Effect of Weight Loss on Myocardial Metabolism and Cardiac Relaxation in Obese Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 05-0523 (201105066); P01HL013851-43 (NIH)
Record Dates: First submitted 2007-12-12; First posted 2007-12-13 (Estimated); Results first posted 2017-05-15 (Actual); Last update posted 2017-05-15 (Actual); Status verified 2017-05

CONDITIONS: Obesity
Keywords: Heart Metabolism; Obesity; Weight loss; Gastric bypass surgery; Diet and exercise
MeSH Terms: conditions — Obesity; Weight Loss; Motor Activity | interventions — Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Diet (Experimental): Participants who received counseling and instruction about weight loss through diet and exercise
  Interventions: Behavioral: Diet
- Gastric bypass surgery (Experimental): Participants who received gastric bypass surgery
  Interventions: Procedure: Gastric bypass surgery

INTERVENTIONS:
Behavioral: Diet — Participants attended 20 group behavioral modification sessions led by a behaviorist, a registered dietician, and a physical therapist. The meal plans ranged from 1200 to 1500 kilocalories per day, depending on subject sex and BMI, and were designed to achieve ≤1% body weight loss/week. Participants completed daily food records, and were taught a variety of weight management skills. The exercise component included strength, flexibility, balance, and endurance instruction, gradually increasing to 30 minutes of exercise 5 days/week.
  Arms: Diet
Procedure: Gastric bypass surgery — The same surgeon performed all bypass procedures using standard techniques. A small (~20 ml) proximal gastric pouch was created by stapling the stomach, and a 75-cm Roux-en-Y limb was constructed by transecting the jejunum distal to the ligament of Treitz, and creating a jejunojejunostomy 75 cm distal to the transection.
  Arms: Gastric bypass surgery

SUMMARY:
Obesity adversely affects myocardial (muscular heart tissue) metabolism, efficiency, and diastolic function. The objective of this study was to determine if weight loss could improve obesity-related myocardial metabolism and efficiency and if these improvements were directly related to improved diastolic function.

DETAILED DESCRIPTION:
This was a prospective, interventional study in obese adults ages 21 to 50 years of age to determine whether weight loss could improve obesity-related myocardial metabolism and efficiency. Two different mechanisms of weight loss were studied: diet and exercise and gastric bypass surgery. Positron emission tomography (PET) was used to quantitate myocardial oxygen consumption (MVO2) and myocardial fatty acid (FA) metabolism. Echocardiography with tissue Doppler imaging was used to quantify cardiac structure, systolic and diastolic function (left ventricular (LV) relaxation (E') and septal ratio (E/E')).

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) > 30 kg/m^2
* Sedentary lifestyle

Exclusion Criteria:

* Body weight >159 kg
* Insulin-requiring diabetes
* Heart failure
* History of coronary artery disease
* Chest pain
* Untreated sleep apnea
* Being an active smoker
* Pregnant, lactating, or postmenopausal

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 51 (Actual)
Dates: Start 2003-06; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Gropler, MD, Principal Investigator — Washington University Medical School
Locations (1):
- Washington University Medical School, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Allison DB, Fontaine KR, Manson JE, Stevens J, VanItallie TB. Annual deaths attributable to obesity in the United States. JAMA. 1999 Oct 27;282(16):1530-8. doi: 10.1001/jama.282.16.1530. PMID 10546692
- [Background] Hu FB, Stampfer MJ, Manson JE, Grodstein F, Colditz GA, Speizer FE, Willett WC. Trends in the incidence of coronary heart disease and changes in diet and lifestyle in women. N Engl J Med. 2000 Aug 24;343(8):530-7. doi: 10.1056/NEJM200008243430802. PMID 10954760
- [Background] Folsom AR, Prineas RJ, Kaye SA, Munger RG. Incidence of hypertension and stroke in relation to body fat distribution and other risk factors in older women. Stroke. 1990 May;21(5):701-6. doi: 10.1161/01.str.21.5.701. PMID 2339449
- [Background] Carey VJ, Walters EE, Colditz GA, Solomon CG, Willett WC, Rosner BA, Speizer FE, Manson JE. Body fat distribution and risk of non-insulin-dependent diabetes mellitus in women. The Nurses' Health Study. Am J Epidemiol. 1997 Apr 1;145(7):614-9. doi: 10.1093/oxfordjournals.aje.a009158. PMID 9098178
- [Result] Lin CH, Kurup S, Herrero P, Schechtman KB, Eagon JC, Klein S, Davila-Roman VG, Stein RI, Dorn GW 2nd, Gropler RJ, Waggoner AD, Peterson LR. Myocardial oxygen consumption change predicts left ventricular relaxation improvement in obese humans after weight loss. Obesity (Silver Spring). 2011 Sep;19(9):1804-12. doi: 10.1038/oby.2011.186. Epub 2011 Jul 7. PMID 21738241
- [Derived] Peterson LR, Saeed IM, McGill JB, Herrero P, Schechtman KB, Gunawardena R, Recklein CL, Coggan AR, DeMoss AJ, Dence CS, Gropler RJ. Sex and type 2 diabetes: obesity-independent effects on left ventricular substrate metabolism and relaxation in humans. Obesity (Silver Spring). 2012 Apr;20(4):802-10. doi: 10.1038/oby.2011.208. Epub 2011 Aug 4. PMID 21818149

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Gastric bypass surgery participants were recruited from the Barnes-Jewish Hospital bariatric surgery center. Diet and exercise participants were recruited from the Volunteer for Health office of Washington University School of Medicine.
Period: Overall Study
Arm/Group | Diet | Gastric Bypass Surgery
Started | 37 | 14
Completed | 20 | 10
Not Completed | 17 | 4
Not completed — Lost to Follow-up | 10 | 4
Not completed — Wanted to do a different diet program | 1 | 0
Not completed — Medication change | 1 | 0
Not completed — Started a new job-- no time for study | 1 | 0
Not completed — Admitted to being a smoker | 1 | 0
Not completed — Refused to do the stress test | 1 | 0
Not completed — Problem with vascular access | 1 | 0
Not completed — Health issues unrelated to the study | 1 | 0

BASELINE CHARACTERISTICS:
Population: Participants who lost 5% of their total body weight following either the diet or gastric bypass surgery interventions
Groups:
- Total: Total of all reporting groups
Arm/Group | Diet | Gastric Bypass Surgery | Total
Number analyzed (Participants) | 20 | 10 | 30
Age, Customized [Count of Participants; unit: Participants]
  ≥ 21 and ≤ 50 years of age | 20 | 10 | 30
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 10 | 22
  Male | 8 | 0 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 20 | 10 | 30
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 0 | 5
  White | 15 | 10 | 25
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 20 | 10 | 30

OUTCOME MEASURES:

1. Primary Outcome: Total Myocardial Oxygen Consumption (MVO2)
Description: The evening before an imaging study, all participants were given a meal containing 12 kcal/kg adjusted body weight (=ideal body weight + ((actual body weight-ideal body weight) x 0.25)). Participants fasted until their imaging studies were completed. Myocardial oxygen consumption (MVO2) was measured using positron emission tomography (PET) following injection of 1-^11C-acetate. Total MVO2 was calculated by multiplying the MVO2 measure by left ventricular weight.
Time Frame: Measured at baseline, 16 months after gastric bypass surgery-induced weight loss, and 8 months after diet-induced weight loss
Population: Participants who lost 5% of their body weight during the study
Measure: Mean (Standard Deviation); unit: µmol/min
Arm/Group | Diet | Gastric Bypass Surgery
Number analyzed (Participants) | 20 | 10
µmol/min
  Baseline | 1064 (318) | 1202 (373)
  Post-intervention | 947 (309) | 835 (232)

2. Primary Outcome: Total Myocardial Fatty Acid (FA) Utilization
Description: The evening before an imaging study, all participants were given a meal containing 12 kcal/kg adjusted body weight (=ideal body weight + ((actual body weight-ideal body weight) x 0.25)). Participants fasted until their imaging studies were completed. Myocardial blood flow was measured using positron emission tomography (PET) following injection of ^30O-water. Myocardial fatty acid (FA) utilization was measured using PET after injection of 1-^11C-palmitate. The calculations that describe the relationship between the different measures of myocardial FA metabolism are: FA utilization/gram = blood flow/gram × FA uptake/gram × [average plasma free FA at the time of the 1-11C-palmitate injection]; FA utilization/gram = FA oxidation/gram + esterification/gram. Total fatty acid utilization was calculated by multiplying the fatty acid utilization rate by left ventricular weight.
Time Frame: as for outcome 1
Population: Participants who lost 5% of their body weight during the study and for whom data are available
Measure: Mean (Standard Deviation); unit: nmol/g/min
Arm/Group | Diet | Gastric Bypass Surgery
Number analyzed (Participants) | 20 | 9
nmol/g/min
  Baseline | 148 (38) | 166 (48)
  Post-intervention | 144 (36) | 148 (79)

3. Primary Outcome: Total Myocardial Fatty Acid (FA) Oxidation
Description: The evening before an imaging study, all participants were given a meal containing 12 kcal/kg adjusted body weight (=ideal body weight + ((actual body weight-ideal body weight) x 0.25)). Participants fasted until their imaging studies were completed. Myocardial fatty acid utilization was measured using positron emission tomography (PET) after injecting 1-^11C-palmitate. Total fatty acid oxidation was calculated by multiplying the fatty acid oxidation rate by left ventricular weight.
Time Frame: as for outcome 1
Population: Participants who lost 5% of their body weight during the study and for whom data are available
Measure: Mean (Standard Deviation); unit: nmol/g/min
Arm/Group | Diet | Gastric Bypass Surgery
Number analyzed (Participants) | 20 | 9
nmol/g/min
  Baseline | 134 (37) | 141 (47)
  Post-intervention | 128 (37) | 127 (50)

4. Secondary Outcome: Left Ventricular (LV) Relaxation (E')
Description: Immediately following MVO2 measurement, complete two-dimensional, M-mode, and Doppler echocardiographic studies were performed using second harmonic imaging. Left ventricular relaxation (E') was measured at the lateral annulus. All reported measurements represent the average of three consecutive cardiac cycles. A single investigator blinded to all clinical parameters evaluated all echocardiograms.
Time Frame: as for outcome 1
Population: Participants who lost 5% of their body weight during the study and for whom data are available
Measure: Mean (Standard Deviation); unit: cm/second
Arm/Group | Diet | Gastric Bypass Surgery
Number analyzed (Participants) | 20 | 9
cm/second
  Baseline | 14.0 (2.7) | 8.2 (1.2)
  Post-intervention | 14.1 (2.2) | 10.4 (1.8)

5. Secondary Outcome: Septal Ratio (E/E')
Description: Immediately following MVO2 measurement, complete two-dimensional, M-mode, and Doppler echocardiographic studies were performed using second harmonic imaging. The early diastolic (E) velocity was measured, left ventricular relaxation (E') was measured at the lateral mitral annulus, and the E/E'(septal) ratio was calculated. All reported measurements represent the average of three consecutive cardiac cycles. A single investigator blinded to all clinical parameters evaluated all echocardiograms. The normal septal ratio from the lateral mitral annulus is <5, a ratio from 5 to 10 is indeterminate, and a ratio of >10 indicates elevated left atrial pressure.
Time Frame: as for outcome 1
Population: Participants who lost 5% of their body weight during the study and for whom data are available
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Diet | Gastric Bypass Surgery
Number analyzed (Participants) | 18 | 7
ratio
  Baseline | 5.9 (1.1) | 12.5 (2.1)
  Post-intervention | 6.1 (1.1) | 8.1 (0.9)

6. Secondary Outcome: Left Ventricular (LV) Mass
Description: Immediately following MVO2 measurement, complete two-dimensional, M-mode, and Doppler echocardiographic study were performed using second harmonic imaging. Left ventricular (LV) mass was measured using the area-length method. All reported measurements represent the average of three consecutive cardiac cycles. A single investigator blinded to all clinical parameters evaluated all echocardiograms.
Time Frame: as for outcome 1
Population: Participants who lost 5% of their body weight during the study and for whom data are available
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | Diet | Gastric Bypass Surgery
Number analyzed (Participants) | 20 | 9
grams
  Baseline | 186 (34) | 180 (24)
  Post-intervention | 186 (32) | 141 (20)

7. Secondary Outcome: Mean Heart Rate
Description: Heart rate was measured at scheduled physical examinations.
Time Frame: as for outcome 1
Population: Participants who lost 5% of their body weight during the study
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Diet | Gastric Bypass Surgery
Number analyzed (Participants) | 20 | 10
beats per minute
  Baseline | 69 (11) | 72 (13)
  Post-intervention | 61 (12) | 65 (17)

8. Secondary Outcome: Mean Arterial Pressure
Description: Mean arterial pressure was measured at scheduled physical examinations.
Time Frame: as for outcome 1
Population: Participants who lost 5% of their body weight during the study
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Diet | Gastric Bypass Surgery
Number analyzed (Participants) | 20 | 10
mm Hg
  Baseline | 89 (9) | 89 (6)
  Post-intervention | 89 (10) | 86 (9)

9. Secondary Outcome: Mean Body Mass Index
Description: Participant weight and height was measured at scheduled physical examinations. Body mass index was calculated as participant body weight in kilograms divided by their height in meters squared.
Time Frame: as for outcome 1
Population: Participants who lost 5% of their body weight during the study
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Diet | Gastric Bypass Surgery
Number analyzed (Participants) | 20 | 10
kg/m^2
  Baseline | 39 (6) | 44 (7)
  Post-intervention | 36 (7) | 29 (5)

10. Secondary Outcome: Mean Total Serum Cholesterol and Triglycerides
Description: Blood testing was conducted at scheduled times during the study. Serum cholesterol and triglycerides were measured by the enzymatic method (Roche Diagnostics).
Time Frame: as for outcome 1
Population: Participants who lost 5% of their body weight during the study
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Diet | Gastric Bypass Surgery
Number analyzed (Participants) | 20 | 10
mg/dl
  Total serum cholesterol, baseline | 182 (38) | 167 (33)
  Total serum cholesterol, post-intervention | 153 (35) | 136 (27)
  Serum triglycerides, baseline | 153 (112) | 168 (90)
  Serum triglycerides, post-intervention | 118 (73) | 72 (21)

11. Secondary Outcome: Mean Homeostasis Model Assessment of Insulin Resistance
Description: The homeostasis model assessment of insulin resistance (HOMA) was used to calculate insulin resistance using the first AM, fasting glucose and insulin levels. Plasma insulin levels were measured by radioimmunoassay, and glucose levels were measured by automated hexokinase assay. A HOMA score of <3 represents normal insulin resistance, a score between 3 and 5 moderate insulin resistance, and a score of 5 or higher represents severe insulin resistance.
Time Frame: as for outcome 1
Population: Participants who lost 5% of their body weight during the study
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Diet | Gastric Bypass Surgery
Number analyzed (Participants) | 20 | 10
units on a scale
  Baseline | 3.8 (2.0) | 5.5 (5.3)
  Post-intervention | 2.7 (1.5) | 0.9 (0.4)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the baseline visit through 8 months for the diet group and through 16 months for the gastric bypass surgery group.
Arm/Group | Diet | Gastric Bypass Surgery
Serious Adverse Events (participants affected / at risk) | 0/37 | 0/14
Other Adverse Events (participants affected / at risk) | 0/37 | 0/14

LIMITATIONS AND CAVEATS:
While this study does show the strength of the relationships between myocardial FA metabolism and MVO2 and relaxation, it does not prove cause and effect, direction of the association, or the potential influence of unmeasured factors.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes